CLINICAL TRIAL: NCT02276313
Title: BIOTRONIK - A Prospective, International, Mulit-centre, Post-market All-comers Registry to Assess the Clinical Performance of the Passeo-18 Lux Paclitaxel Releasing Balloon Catheter in Infrainguinal Arteries - III
Brief Title: BIOLUX P-III All-Comers Passeo-18 Lux Registry
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1211
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Atherosclerosis; Peripheral Artery Disease
Keywords: Peripheral; Infrainguinal; Drug Releasing Balloon; Drug Eluting Balloon
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Passeo-18 Lux — Endovascular Therapy

SUMMARY:
BIOLUX P-III is a prospective, international, multi-centre, postmarket all-comers registry to collect clinical performance data on the Passeo-18 Lux paclitaxel releasing balloon catheter in the treatment of atherosclerotic disease of the infrainguinal arteries.

DETAILED DESCRIPTION:
The Passeo-18 LUX Paclitaxel Releasing BalloonCatheter is a novel drug-releasing balloon that received CE-mark in January 2014. Its safety and efficacy has been investigated in two randomized First-in-Man trials in patients with stenosis or occlusion of the femoropopliteal (BIOLUX P-I) and infrapopliteal (BIOLUX P-II) arteries when compared to an uncoated device.

The purpose of the BIOLUX P-III all-comers registry is to collect short and long-term clinical performance data on the Passeo-18 Lux DRB in the treatment of atherosclerotic disease in the infrainguinal arteries in an all-comers patient population in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum age as required by local regulations
* Subject must be willing to sign a Patient Data Release Form or Patient Informed Consent where applicable
* Lesion(s) in the infrainguinal arteries suitable for endovascular treatment treated with or scheduled to be treated with the Passeo-18 Lux drug releasing balloon

Exclusion Criteria:

* Life expectancy ≤ 1 year
* Subject is currently participating in another investigational drug or device study that has not reached ist primary endpoint yet
* Subject is pregnant or planning to become pregnant during the course of the study
* Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion in the absence of flow limiting dissections or perforations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from an all-comers patient population with all subjects requiring infrainguinal revascularization with the Passeo-18 Lux DRB.
Sampling Method: Non-Probability Sample
Enrollment: 880 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events (MAE) | 6 months
  A composite of freedom from device- and procedure-related mortality through 30 days, freedom from major target limb amputation and clinically driven target lesion revascularization (TLR) within 6 months post-index procedure.
Freedom from clinically-driven Target Lesion Revascularization (TLR) | 12 months

SECONDARY OUTCOMES:
Freedom from clinically-driven TLR | 6 and 24 months
Freedom from clinically-driven Target Vessel Revascularization (TVR) | 6 and 24 months
Primary patency | 12 and 24 months
Freedom from MAE | 12 and 24 months
Change in mean Ankle Brachial Index | 6, 12 and 24 months
Amputation-free survival | 6, 12 and 24 months
Patient-reported outcomes assessment: Pain score, Walking Impairment Questionnaire | 6, 12 and 24 months
Clinical Success: Improvement in Rutherford classification compared to the pre-procedure Rutherford classification | 6, 12 and 24 months
Device success | Day 0
  Successful delivery, inflation, deflation, and retrieval of the Passeo-18 Lux DRB.
Technical success | Day 0
  Successful completion of the endovascular procedure and immediate morphological success with ≤ 50% residual diameter reduction of the treated lesion as determined by visual estimation
Procedural success | Participants will be followed for the duration of hospital stay, an expected average of 1-2 days
  Procedural success is technical and device success without the occurrence of any major adverse events during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — RoMed Klinikum Rosenheim
Locations (45):
- Australia (5):
  - Cairns Hospital, Cairns
  - Lake Macquarie Private Hospital, Gateshead
  - Geelong University Hospital, Geelong
  - Hollywood Hospital, Nedlands
  - The Townsville Hospital, Townsville
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Department Radiologie, Universitätsklinik für Radiodiagnostik, Innsbruck
- Belgium (4):
  - UCL St. Luc, Brussels
  - UZ Leuven, Leuven
  - CHR de la Citadelle, Liège
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
- Kolding Hospital, Kolding, Denmark
- Tampereen Yliopiostollinen Keskussariaaia, Tampere, Finland
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Clinique Pasteur Essey Les Nancy, Essey-lès-Nancy
  - CHU de Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon
- Germany (10):
  - Klinikum Arnsberg, Karolinenhospital, Arnsberg
  - Department of Angiology at Universitats- Herzzentrum Freiburg, Bad Krozingen
  - Gemeinschaftspraxis für Radiologie, Berlin
  - Sank Gertrauden-Krankenhaus, Berlin
  - Universitätsklinikum Giessen und Marburg GmbH, Giessen
  - Herz- und Gefässzentrum Göttingen, Göttingen
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Kliniken München Pasing-Perlach GmbH, München Pasing
  - RoMed Klinikum Rosenheim, Rosenheim
- Italy (2):
  - Ospedale San Giovanni di Dio, Florence
  - Policlinico San Donato, San Donato Milanese
- P.Stradins Clinical University Hospital, Institute of Diagnostic, Riga, Latvia
- Institute Jantung Negara, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - Saint Elisabeth Hospital, Tilburg
- Hospital Garcia de Orta, Almada, Portugal
- Singapore (3):
  - Changi General Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Institute of Cardiovascular diseases Kosice, Dpt. of Angiology, Košice, Slovakia
- Spain (4):
  - Hospital. Universitario Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Severo Ochoa, Madrid
- Switzerland (3):
  - Centre Hopsitalier Universitaire Vaudois, Lausanne
  - Ospedale Regionale di Lugano, Lugano
  - KS Winterthur, Winterthur

REFERENCES:
- [Derived] Dodd JE, Hanna J, Brodmann M, Golledge J, Zeller T, Moscovic M, Dahm J, Troisi N, Tepe G, Wong J, Ward NC, Mwipatayi BP. Outcomes of drug-coated balloon angioplasty in patients with dyslipidemia in the BIOLUX P-III registry: A subgroup analysis. Vascular. 2025 Dec;33(6):1288-1303. doi: 10.1177/17085381241275795. Epub 2024 Aug 19. PMID 39158589
- [Derived] Barry IP, Macarulay R, Brodmann M, Zeller T, Moscovic M, Dahm J, Troisi N, Tepe G, Wong J, Mwipatayi BP; BIOLUX P-III Global Registry Investigators. Sex-Related Outcomes Following Drug Balloon Angioplasty in Patients from the BIOLUX P-III Registry: A Subgroup Analysis. Cardiovasc Intervent Radiol. 2022 Jul;45(7):918-928. doi: 10.1007/s00270-022-03135-w. Epub 2022 Apr 20. PMID 35445317
- [Derived] Mwipatayi BP, Barry IP, Brodmann M, Zeller T, Varcoe RL, Moscovic M, Chian JWC, Christensen JK, Yahaya SA, Oshin OA, Tepe G; BIOLUX P-III Global Registry Investigators. Twenty-Four-Month Outcomes of Drug-Coated Balloon in Diabetic Patients in the BIOLUX P-III Registry: A Subgroup Analysis. Ann Vasc Surg. 2021 Aug;75:237-252. doi: 10.1016/j.avsg.2021.02.050. Epub 2021 Apr 5. PMID 33831519
- [Derived] Tepe G, Zeller T, Moscovic M, Corpataux JM, Christensen JK, Keirse K, Nano G, Schroeder H, Binkert CA, Brodmann M. Paclitaxel-Coated Balloon Angioplasty for the Treatment of Infrainguinal Arteries: 24-Month Outcomes in the Full Cohort of BIOLUX P-III Global Registry. Cardiovasc Intervent Radiol. 2021 Feb;44(2):207-217. doi: 10.1007/s00270-020-02663-7. Epub 2020 Oct 20. PMID 33083853
- [Derived] Tepe G, Wang J, Corpataux JM, Pua U, Binkert CA, Moscovic M, Ghotbi R, Keirse K, Robertson D, Brodmann M. BIOLUX P-III Passeo-18 Lux All-Comers Registry: 24-Month Results in Below-the-Knee Arteries. Cardiovasc Intervent Radiol. 2021 Jan;44(1):10-18. doi: 10.1007/s00270-020-02586-3. Epub 2020 Sep 22. PMID 32964317
- [Derived] Tepe G, Zeller T, Moscovic M, Corpataux JM, Christensen JK, Keirse K, Nano G, Schroeder H, Binkert CA, Brodmann M. Paclitaxel-Coated Balloon for the Treatment of Infrainguinal Disease: 12-Month Outcomes in the All-Comers Cohort of BIOLUX P-III Global Registry. J Endovasc Ther. 2020 Apr;27(2):304-315. doi: 10.1177/1526602819898804. Epub 2020 Jan 28. PMID 31989855